CLINICAL TRIAL: NCT06152159
Title: Postpartum Experience by the Second Parent
Acronym: PostPartum2ndP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_018_PostPartum-2ndP
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Postpartum Experience
Keywords: postpartum experience; second parent
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The second parent of a child: The second parent of a child born since minimum 3 months and maximum 6 months.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Data collection

SUMMARY:
Many studies have been performed on mothers and their postnatal experiences. Unfortunately, studies about the second parent are very rare. Second parent is yet an essential figure in the parent-child triad and a real support for the mother.

The postpartum period is a time of intense restructuring and upheaval, both physically and psychologically. Studies have shown that almost 13% of fathers suffer from depression.

DETAILED DESCRIPTION:
The main objective is to describe the postpartum experience of the second parent.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Second parent of a child born living for at least 3 months and at most 6 months
* Major
* Agreeing to participate in the study

Exclusion Criteria:

* Minors
* Protected by law (guardianship, curatorship, safeguarding of justice)
* Not agreeing to participate in this study
* Parents of stillborn children
* Refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The second parent of a child born since minimum 3 months and maximum 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Experience of the postpartum by the second parent | Day 0
  This experience of the postpartum by the second parent will be evaluated by a Likert scale with 5 proposals:
  Very good experience/ Good experience/ Lived/neutral/ Bad experience/ Very bad experience

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided